CLINICAL TRIAL: NCT00000454
Title: Field Study of Smoking Cessation in Alcoholism Treatment
Brief Title: Smoking Cessation in Alcoholism Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NIAAACOO11197; R01AA011197 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Alcoholism; Smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: nicotine replacement patch

SUMMARY:
This study is designed to increase understanding of the processes that affect the treatment outcome of individuals with both alcohol and nicotine dependence. Treatment outcome methodology will be combined with a computerized self-monitoring methodology to examine the extent to which smoking serves as a cue for alcohol craving and/or as a response to alcohol craving in treated alcoholics. Subjects will be veterans participating in the Substance Abuse Day Programs at the Newington and West Haven campuses of the VA Connecticut Healthcare System. Nonveteran women will be recruited from the community and enrolled in the day program. Subjects will be randomly assigned to one of the following two conditions: (1) intensive smoking cessation therapy (counseling plus nicotine replacement using nicotine patches) concurrent with alcohol treatment, or (2) brief smoking cessation advice concurrent with alcohol treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence within the past three months, and criteria for nicotine dependence.
* Smoking at least 10 or more cigarettes per day for the past year.
* Seeking treatment for both alcohol and nicotine dependence.
* Minimum 1 week of alcohol abstinence and substance abuse day treatment attendance.
* Willing to provide names of two individuals who can help locate the subject at follow-up.
* Willing to provide name of one individual who can provide collateral information about alcohol and tobacco use.

Exclusion Criteria:

* Other substance use disorder meeting criteria for dependence.
* Acute medical or psychiatric disorder requiring inpatient treatment.
* Taking medications known to influence alcohol urges (naltrexone, disulfiram).
* Medical problems that would contraindicate nicotine patch use.
* Allergy or hypersensitivity to nicotine or to adhesives used in transdermal delivery systems.
* Use of other nicotine products such as cigars, pipes, or smokeless tobacco.
* Severe generalized skin disorder.
* Myocardial infarction within 3 months prior to study entry.
* Unstable angina.
* Pregnant or lactating females, or females who are not practicing a medically accepted form of contraception.
* Impaired vision or hearing which would interfere with using a hand-held computer.
* Reading ability below fifth grade level.
* Lack of reliable transportation to the treatment site, or living more than 1 hour from treatment site.
* Homeless or unstable residence.
* Plan for future admission to residential treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- Substance Abuse Treatment Center, VA Medical Center, West Haven, Connecticut, United States

REFERENCES:
- [Result] Cooney NL, Litt MD, Cooney JL, Pilkey DT, Steinberg HR, Oncken CA. Concurrent brief versus intensive smoking intervention during alcohol dependence treatment. Psychol Addict Behav. 2007 Dec;21(4):570-5. doi: 10.1037/0893-164X.21.4.570. PMID 18072840
- [Result] Cooney NL, Litt MD, Cooney JL, Pilkey DT, Steinberg HR, Oncken CA. Alcohol and tobacco cessation in alcohol-dependent smokers: analysis of real-time reports. Psychol Addict Behav. 2007 Sep;21(3):277-86. doi: 10.1037/0893-164X.21.3.277. PMID 17874878